CLINICAL TRIAL: NCT04353518
Title: A Randomized, Double-blind, Two Arm, Placebo Controlled Clinical Trial to Evaluate the Efficacy and Safety of Mycobacterium w in Preventing COVID-19 in Subjects at Risk of Getting Infected With COVID-19.
Brief Title: Clinical Trial to Evaluate Mycobacterium w in Preventing COVID-19 in Subjects at Risk of Getting Infected With COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cadila Pharnmaceuticals (Industry)
Collaborators: Council of Scientific and Industrial Research, India (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRSC20005
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, two arms, placebo controlled, clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suspension of Mw (Experimental): Intradermal suspension of Mw will be administered in two divided doses:
  Dose 1 at Day 0: 0.2 ml (0.1 ml x 2 injection) of intradermal Mw in two divided dose.
  Dose 2 at Day 15 after the first dose: 0.1 ml injection of intradermal Mw administered.
  Interventions: Drug: Suspension of heat killed (autoclaved) Mycobacterium w
- Placebo (Placebo Comparator): Placebo will be administered in two divided doses:
  Dose 1 at Day 0: 0.2 ml (0.1 ml x 2 injection) of intradermal placebo in two divided dose.
  Dose 2 at Day 15 after the first dose: 0.1 ml injection of intradermal placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Suspension of heat killed (autoclaved) Mycobacterium w — Subjects randomized to Test arm will receive intraderma Mw in divided doses at least 2 cm away from first injection site in the deltoid region.
  Arms: Suspension of Mw
Other: Placebo — Subjects randomized to placebo arm will receive intraderma Placebo in divided doses at least 2 cm away from first injection site in the deltoid region.
  Arms: Placebo

SUMMARY:
This clinical trial is a randomized, blinded, two arms, placebo controlled, clinical trial to evaluate the safety and efficacy of Mycobacterium w in combination with standard care as per hospital practice to prevent COVID 19 in subjects at risk of getting infected with COVID 19.

DETAILED DESCRIPTION:
Approximately eligible 4000 subjects who are at risk of getting infected with COVID-19 (i.e. person living in same household as COVID-19 patients / healthcare workers providing direct care to COVID-19 patients) will be enrolled in to the study after due consent and based on the eligibility criteria.

Initially, 400 subjects at risk of getting infected with COVID-19 will be enrolled in the study and randomized in 1:1 ratio to receive either Mw (n=200) or placebo (n=200). After the interim analysis from the data of these 400 subjects for safety and efficacy and based on review and recommendations from DSMB / MC, modification in study design, objective or sample size will be considered.

Study duration for each subject will be of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of either gender, age ≥ 18 years, with recent history of close contact with COVID-19 patients.
* Subjects with SARS Cov 2 negative test (ICMR approved test kit) at screening visit.
* Female subject who are currently using reliable methods of contraception (barrier methods and intrauterine contraceptive device), with a negative urine pregnancy test during screening and agree to informed compliance of contraceptive method until at least months post-dosing.
* The subject must be able and willing to comply with the study protocol, available and willing to complete all the study assessments and must have signed an Informed Consent Form.

Exclusion Criteria:

* Any febrile illness with oral temperature > 100°F within 3 days prior to randomization.
* Subject with past history of COVID-19 infection.
* Pregnant and / or lactating female subjects.
* Presence of any illness requiring hospital referral.
* Any confirmed or suspected immune-deficient condition based on medical history and physical examination and a family history of congenital or hereditary immunodeficiency or Individuals on immunosuppressant's as Azathioprine, Cyclosporine, Mycophenolate etc.
* History of allergic reactions or anaphylaxis to Mw or its component.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of subject acquiring COVID-19 infection | From first dosing to week 1, week 2, week 4, week 8 or at any time during the study till 8 week post first dosing..
  To compare proportion of subjects acquiring COVID-19 infection between two arms over the time till 8 weeks from administration of 1st dose

SECONDARY OUTCOMES:
Incidence of Adverse Event and Serious Adverse Event (safety and tolerability) | Till 8 weeks
  Any AE / SAE observed during the study.
Number of subject developing Upper Respiratory Tract Infection (URTI) symptoms | From first dosing to week 1, week 2, week 4, week 8 or at any time during the study till 8 week post first dosing.
  Whether administration of Mw prevents development of Upper Respiratory Tract Infection (URTI) symptoms in close contacts of COVID-19 patients.
Number of subject developing severe COVID-19 infection based on ordinal scale | From first dosing to week 1, week 2, week 4, week 8 or at any time during the study till 8 week post first dosing
  Whether administration of Mw prevents development of severe COVID-19 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Avhad, MBBS, Study Chair — Cadila Pharmaceuticals Limited
Locations (3):
- India (3):
  - All India Institute of Medical Sciences, Bhopal, Bhopal, Madhya Pradesh
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - All lndia Institute of Medical Science, Delhi, Delhi

IPD SHARING:
Plan to Share IPD: No